CLINICAL TRIAL: NCT04557046
Title: A Multicenter COVID-19 Study Conducted to Evaluate the Performance of the LumiraDx SARS-CoV-2 Ag Test at Point of Care Testing Sites
Brief Title: Performance Evaluation of LumiraDx COVID-19 (SARS-CoV-2) Ag Test
Acronym: ASPIRE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: LumiraDx UK Limited (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: S-CLIN-PROT-00032
Record Dates: First submitted 2020-09-17; First posted 2020-09-21 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-12

CONDITIONS: Covid19
Keywords: POC; SARS-CoV-2; Antigen
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Subject are asked to provide nasal swab or nasopharyngeal swab and saliva samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (5):
- Group A: Sample Collection (Other): Nasal Swab and Saliva Sample Collection
  Interventions: Diagnostic Test: Nasal Swab; Diagnostic Test: Saliva specimen
- Group B: Sample Collection (Other): Nasal swab, Capillary Blood (from fingerstick) and Saliva Collection
  Interventions: Diagnostic Test: Nasal Swab; Diagnostic Test: Fingerstick; Diagnostic Test: Saliva specimen
- Group C: Sample Collection (Other): Nasal Swab, Throat Swab and Saliva Sample Collection
  Interventions: Diagnostic Test: Nasal Swab; Diagnostic Test: Throat swab; Diagnostic Test: Saliva specimen
- Group D: Sample Collection (Other): Nasopharyngeal Swab and Saliva Sample Collection
  Interventions: Diagnostic Test: Nasopharyngeal swab; Diagnostic Test: Saliva specimen
- Group E: Sample Collection (Other): Nasal swab
  Interventions: Diagnostic Test: Nasal Swab

INTERVENTIONS:
Diagnostic Test: Nasal Swab — Collection of one more nasal swabs
  Arms: Group A: Sample Collection; Group B: Sample Collection; Group C: Sample Collection; Group E: Sample Collection
Diagnostic Test: Nasopharyngeal swab — Collection of one more nasopharyngeal swabs
  Arms: Group D: Sample Collection
Diagnostic Test: Throat swab — Collection of one more throat swabs
  Arms: Group C: Sample Collection
Diagnostic Test: Fingerstick — Collection of capillary blood from one or more fingersticks
  Arms: Group B: Sample Collection
Diagnostic Test: Saliva specimen — Collection of free drool
  Arms: Group A: Sample Collection; Group B: Sample Collection; Group C: Sample Collection; Group D: Sample Collection

SUMMARY:
Performance of the LumiraDx SARS-CoV-2 Ag assay will be assessed by comparison to a reference method.

DETAILED DESCRIPTION:
The study is a prospective, multi-center study. One (1) reference laboratory and approximately six (6) geographically diverse POC (Point of Care) locations (e.g. physician office laboratories, urgent cares, emergency departments, outpatient clinics, drive through testing sites or research centers) in the U.S. will participate in the study. Testing in the reference laboratory will be performed by trained laboratory personnel. Testing at the POC sites will be performed by non-laboratory health professionals who are representative of typical intended use operators (e.g. nurses, physician assistants, medical assistants, etc.). Each site will have a minimum of one (1) untrained intended use operator who will perform testing under this protocol.

A subject's participation in this study will consist of a single visit. Following completion of the informed consent process and a review of Inclusion/Exclusion criteria to determine eligibility, each subject will receive a unique study identification number.

Subjects will have nasopharyngeal or nasal or throat swabs collected. Capillary blood may be collected alongside nasal swabs. Saliva samples may also be collected. Specimens will be obtained from each subject enrolled using standard collection methods.

The LumiraDx SARS-CoV-2 Ag Test will be performed at POC sites by intended use operators (e.g. nurses, physician assistants, medical assistants, etc.). Each site will have a minimum of one (1) untrained intended use operator who will perform testing under this protocol.

The LumiraDx SARS-CoV-2 Ag Test will be performed at the site on the same day as the date of collection using one swab for each subject enrolled. A central laboratory will perform reference testing.

Positive Percent Agreement (PPA) and Negative Percent Agreement (NPA) will be estimated for the LumiraDx SARS-CoV-2 Ag Test results as compared with the reference Test.

A minimum of thirty (30) positive SARS-CoV-2 are required, but it is likely because of the prevalence of SARS-CoV-2 in the population, that a greater number of negatives will be obtained during the prospective collection of positive samples; therefore, approximately four-hundred (400) subjects will be enrolled. A minimum of thirty (30) negative samples are required.

ELIGIBILITY:
Inclusion Criteria:

* 1. The subject may be of any age and either sex.
* 2. Preliminary assessment of the subject by the Investigator/designee should be suggestive of COVID-19 at the time of the study visit. The subject must present as symptomatic, meaning they have exhibited one or more of the following signs and symptoms for eligibility: fever, cough, shortness of breath, difficulty breathing, muscle pain, headache, sore throat, chills, repeated shaking with chills, new loss of taste or smell. The onset of these symptoms will be recorded.

or The subject must have a documented SARS-CoV-2 PCR test in the past 48 hours.

* 3. Written informed consent must be obtained prior to study enrollment.

  1. A subject who is eighteen (18) years or older must be willing to give written informed consent and must agree to comply with study procedures.
  2. The Legal Guardian or Legal Authorized Representative of a subject who is under the age of eighteen (18) must give written informed consent and agree to comply with study procedures. Active written assent should be obtained from children of appropriate intellectual age (as defined by the IRB).

Exclusion Criteria:

* 1. The subject underwent a nasal wash/aspirate as part of standard of care testing during this study visit.
* 2. The subject is currently receiving or has received within the past thirty (30) days of the study visit an experimental biologic, drug, or device including either treatment or therapy.
* 3. The subject has previously participated in this research study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1134 (Actual)
Dates: Start 2020-06-26 (Actual); Primary Completion 2021-03-24 (Actual); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
Performance Evaluation | 4 months
  Evaluation of performance of the device versus a reference method using standard qualitative comparison techniques (Percent Agreement)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Chappel, Principal Investigator — Chappel Group; Robert Rosen, Principal Investigator — Ardmore Family Practice; Andre Gvozden, Principal Investigator — Gvozden Pediatrics; Madhavi Ampajwala, Principal Investigator — Village Health Partners; Edward Zissman, Principal Investigator — Pediatric Associates of Altamonte Springs; Melanie Hoppers, Principal Investigator — Physicians Quality Care of Jackson; Kimberley Henderson, Principal Investigator — Good Samaritan Minute Clinic
Locations (7):
- United States (7):
  - Children's Pediatric Associates of Altamonte Springs, Altamonte Springs, Florida
  - Chappel Group, Kissimmee, Florida
  - Good Samaritan Minute Clinic, Georgia Tech, Atlanta, Georgia
  - Gvozden Pediatrics, Millersville, Maryland
  - Ardmore Family Practice, Winston-Salem, North Carolina
  - Physicians Quality Care of Jackson, Jackson, Tennessee
  - Village Health Partners, Plano, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ellis JE, Guest P, Lawson V, Loecherbach J, Lindner N, McCulloch A. Performance Evaluation of the Microfluidic Antigen LumiraDx SARS-CoV-2 and Flu A/B Test in Diagnosing COVID-19 and Influenza in Patients with Respiratory Symptoms. Infect Dis Ther. 2022 Dec;11(6):2099-2109. doi: 10.1007/s40121-022-00696-8. Epub 2022 Sep 24. PMID 36152227
- [Derived] Drain PK, Ampajwala M, Chappel C, Gvozden AB, Hoppers M, Wang M, Rosen R, Young S, Zissman E, Montano M. A Rapid, High-Sensitivity SARS-CoV-2 Nucleocapsid Immunoassay to Aid Diagnosis of Acute COVID-19 at the Point of Care: A Clinical Performance Study. Infect Dis Ther. 2021 Jun;10(2):753-761. doi: 10.1007/s40121-021-00413-x. Epub 2021 Feb 24. PMID 33629225